CLINICAL TRIAL: NCT01386229
Title: A Comparison of Etomidate and Ketamine for Anesthesia Induction in Coronary Artery Bypass Graft Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Özgür Kömürcü, Baskent University, Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KA-10-114
Record Dates: First submitted 2011-06-21; First posted 2011-07-01 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Coronary Artery Bypass Surgery
Keywords: hemodynamic stability; etomidate; ketamine; coronary artery bypass surgery after induction of anesthesia, hemodynamic stability
MeSH Terms: interventions — Ketamine; Etomidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Active Comparator)
  Interventions: Drug: Ketamine
- Etomidate (Active Comparator)
  Interventions: Drug: Etomidate

INTERVENTIONS:
Drug: Ketamine — During standard anesthesia induction with fentanyl and midazolam, ketamine 2 mg/kg IV will be administered
  Arms: Ketamine
Drug: Etomidate — During standard anesthesia induction with fentanyl and midazolam, etomidate 3 mg/kg IV will be administered
  Arms: Etomidate

SUMMARY:
The aim of this study is to determine whether ketamine is an acceptable alternative to etomidate for anesthesia induction in coronary artery bypass graft surgery in terms of hemodynamic stability and also to compare these agents regarding their effect on adrenal gland steroid synthesis in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective coronary artery bypass graft surgery with cardiopulmonary bypass
* Patient's written informed consent for study participation
* Ejection fraction ≥ 35%

Exclusion Criteria:

* Allergy to study drugs
* Redo surgery

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
A more than 15% change in mean arterial pressure and heart rate after anesthesia induction | For 60 minutes after anesthesia induction

SECONDARY OUTCOMES:
Adrenal gland steroid synthesis suppression | 24 hours and 5 days after study drug administration
  A less than 9 microgram/dl increase in serum cortisol after stimulation with adrenocorticotropic hormone

CONTACTS AND LOCATIONS:
Overall Officials: Özgür Kömürcü, Principal Investigator — Baskent University, Faculty of Medicine
Locations (1):
- Baskent University, Faculty of Medicine, Ankara, Çankaya, Turkey (Türkiye)